CLINICAL TRIAL: NCT01368406
Title: Efficacy of a Non-pharmacological Intervention for Weight Gain Management for Patients With Schizophrenia: Multicentric, Randomized Clinical Trial
Brief Title: Lifestyle Intervention for Weight Gain Management for Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Cecilia Attux, principal investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007/00464-6
Record Dates: First submitted 2011-05-17; First posted 2011-06-08 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-04

CONDITIONS: Schizophrenia; Obesity
Keywords: schizophrenia; weight gain; intervention
MeSH Terms: conditions — Schizophrenia; Obesity; Weight Gain | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- wellness program (Experimental): 12-week weight management intervention in patients with severe mental disorders. In the 1-hour weekly group sessions topics like dietary choices, lifestyle, physical activity and self-esteem were discussed with outpatients and their relatives
  Interventions: Behavioral: wellness program
- treatment as usual (No Intervention): patients were on regular visits on psychiatrist

INTERVENTIONS:
Behavioral: wellness program — 12-week weight management intervention in patients with severe mental disorders. In the 1-hour weekly group sessions topics like dietary choices, lifestyle, physical activity and self-esteem were discussed with outpatients and their relatives
  Other Names: brazilian wellness program
  Arms: wellness program

SUMMARY:
The aims of this study were to evaluate the efficacy of an intervention for weight gain management for patients from schizophrenia spectrum compared to treatment as usual (TAU), and to evaluate the effects of this program on metabolic profile, symptoms and quality of life.

DETAILED DESCRIPTION:
The study took place on four institutions: Schizophrenia Program (PROESQ- Universidade Federal de São Paulo), Schizophrenia Program of Institute of Psychiatry PROJESQ (Universidade de São Paulo), CAISM (Centro de Atenção Integrada à Saúde Mental) from Irmandade Santa Casa de Misericórdia de São Paulo, and CAPS Luiz da Rocha Cerqueira, all in the city of São Paulo. Participants were randomly assigned to an intervention group or a standard care group using table of randomization from web site www.randomization.com. The patients' weights were recorded monthly. All patients were weighed in the morning, on the same scale, without shoes, with the individuals wearing light clothes. Waist was considered at the level of the navel. Measures were collected by the same investigator in all assessments. Body mass index (BMI) was calculated as the weight in kilograms divided by the square of the height in meters. The investigators recorded sociodemographic data, clinical data and physical exam (weight, height, BMI, waist circumference and blood pressure). Patients were diagnosed as having schizophrenia by the SCID-P (REF). Severity of the disease was assessed using PANSS, Calgary Depression Scale, CGI-S and CGI-I. GAF, ILSS-BR, and he following self-rated scales: WHOQoL-BREF, Rosenberg self-esteem scale, IPAQ, DINE and Fagerstrom were used to evaluate functionality (GAF), independent living skills (ILSS-BR), quality of life (WHOQoL-BREF), self esteem (Rosenberg self-esteem scale), physical activity (IPAQ- short version), fat and fibers ingestion (DINE), and smoking (Fagerstrom). Raters were kept blind for patient's treatment condition. Fasting glucose, total cholesterol, HDL, LDL, triglycerides, insulin, and HOMA-IR index were assessed at baseline, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were between 18 and 65 years of age,
* were on an antipsychotic medication,
* were asymptomatic (PANSS ≤ 60),
* had outpatient status and a DSM-IV diagnosis of schizophrenia,
* schizoaffective disorder or other psychosis, and
* presented some interest on themes of program.

Exclusion Criteria:

* a history of diabetes mellitus,
* eating disorders (anorexia and bulimia),
* drug or alcohol abuse,
* and an acute psychotic state in need of intensive management.
* There was no use of medication for weight control for the subjects during the intervention and follow-up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Bressan, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (4):
- Brazil (4):
  - Schizophrenia Program (PROESQ), São Paulo, São Paulo
  - Caps Luiz da Rocha Cerqueira, São Paulo, São Paulo
  - Centro de Atenção Integrada à Saúde Mental (CAISM), São Paulo, São Paulo
  - Schizophrenia Program of Institute of Psychiatry PROJESQ, São Paulo, São Paulo

REFERENCES:
- [Derived] Attux C, Martini LC, Elkis H, Tamai S, Freirias A, Camargo Md, Mateus MD, Mari Jde J, Reis AF, Bressan RA. A 6-month randomized controlled trial to test the efficacy of a lifestyle intervention for weight gain management in schizophrenia. BMC Psychiatry. 2013 Feb 18;13:60. doi: 10.1186/1471-244X-13-60. PMID 23418863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were drawn from: a) the Schizophrenia Program- Universidade Federal de São Paulo); b) the Schizophrenia Program of Institute of Psychiatry PROJESQ (Universidade de São Paulo); c) the CAISM (Centro de Atenção Integrada à Saúde Mental) from Irmandade Santa Casa de São Paulo; and d) the Community Psychosocial Center Luiz da Rocha Cerqueira.
Groups:
- Treatment as Usual: treatment as usual received by the patients
Period: Overall Study
Arm/Group | Wellness Program | Treatment as Usual
Started | 81 | 79
Completed | 60 | 66
Not Completed | 21 | 13
Not completed — Lost to Follow-up | 8 | 4
Not completed — Withdrawal by Subject | 8 | 4
Not completed — relapse of the disease | 3 | 2
Not completed — started working | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wellness Program | Treatment as Usual | Total
Number analyzed (Participants) | 81 | 79 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 79 | 160
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.2 (9.9) | 38.3 (10.7) | 37.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 50 | 46 | 96
Region of Enrollment [Number; unit: participants]
  Brazil | 81 | 79 | 160

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight From Baseline to Endpoint
Description: All patients were weighed in the morning, on the same scale, without shoes, with the individuals wearing light clothes.Measures were collected by the same investigator in all assessments.
Time Frame: baseline, 3-month
Measure: Mean (95% Confidence Interval); unit: kg
Groups:
- Wellness Program: lifestyle intervention for 12 weeks
Arm/Group | Wellness Program | Treatment as Usual
Number analyzed (Participants) | 81 | 79
kg | 0.48 [-0.65 to 1.13] | 0.48 (17.8) [0.13 to 0.83]
Statistical Analysis 1: Comparison: Wellness Program; Test type: Superiority or Other; p = 0.055, t-test, 2 sided; t test for independent samples; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.65 to 1.13]
Statistical Analysis 2: Comparison: Treatment as Usual; Test type: Superiority or Other; p = 0.055, t-test, 2 sided; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [0.13 to 0.83]

ADVERSE EVENTS:
Time Frame: Although the intervention lasted 3 months, the study was enrolled during a 3 year period, so we could observe adverse events during this time
Arm/Group | Wellness Program | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/79
Other Adverse Events (participants affected / at risk) | 0/81 | 0/79

LIMITATIONS AND CAVEATS:
short duration of the intervention (12 weeks) and duration of follow up. This lifestyle intervention was previously conducted in all sites that participated of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No